CLINICAL TRIAL: NCT01560572
Title: Steroid Free Immunosuppression or Calcineurin Inhibitor Minimization After Basiliximab Induction Therapy in Kidney Transplantation: Comparison With a Standard Quadruple Immunosuppressive Regimen
Acronym: Allegro
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Leiden University Medical Center (Other); Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, J.S.F. Sanders, principal investigator, University Medical Center Groningen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Allegro
Record Dates: First submitted 2011-12-21; First posted 2012-03-22 (Estimated); Last update posted 2022-01-11 (Actual); Status verified 2021-12

CONDITIONS: Renal Insufficiency; Kidney Transplantation
Keywords: kidney transplantation; immunosuppression; steroids; tacrolimus OD
MeSH Terms: conditions — Renal Insufficiency | interventions — Mycophenolic Acid; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- standard immunosuupression (Active Comparator): triple maintenance immunosuppression with tacrolimus OD (maintenance 6-10 ng/ml), mycophenolic acid 2 dd 540mg and prednisolone 7.5 mg
  Interventions: Drug: tacrolimus OD, mycophenolic acid, prednisolone
- steroidfree (Experimental): maintenance immunosuppression with tacrolimus OD (target range 6-10 ng/ml), mycophenolic acid (2 dd 540 mg)
  Interventions: Drug: tacrolimus OD, mycophenolic acid, prednisolone
- low dose tacrolimus (Experimental): triple maintenance immunosuppression with tacrolimus OD (maintenance 6-10 ng/ml), mycophenolic acid 2 dd 540mg and prednisolone 7.5 mg. After 6 months lowering of tacrolimus OD maintenance 3-5 ng/ml
  Interventions: Drug: tacrolimus OD, mycophenolic acid, prednisolone

INTERVENTIONS:
Drug: tacrolimus OD, mycophenolic acid, prednisolone — tacrolimus maintenance 6-10 ng/ml, in the low dose tacrolimus group after 6 months fixed dose reduction of 50% tacrolimus through levels will be 3-5 ng/ml mycophenolic acid 2 dd 720mg, after 2 weeks reduced to 2 dd 540 mg in all groups methylprednisolone 500, 250, 125 mg on day 0, 1, and 2 in all groups prednisolone 1 dd 10 mg, and from week 6 prednisolone 7.5 mg in the standard immunosuppression and low dose tacrolimus group No prednisolone will be given the steroid free group
  Other Names: advagraf, mycophenolic acid

SUMMARY:
A prospective, open, randomized trial, in which the investigators aim to achieve optimal immunosuppression after renal renal transplantation with maximal reduction of side effects, especially of vascular injury, chronic allograft nephropathy, osteoporosis and malignancies. Immunosuppression without steroids and CNI minimization is compared to standard immunosuppression, consisting of tacrolimus OD, mycophenolic acid and corticosteroids.

DETAILED DESCRIPTION:
Before transplantation 300 patients will be randomized 1:1:1 in three groups. Group 1 will be treated with basiliximab induction and a three day course of steroids followed by a steroid free maintenance regimen consisting of standard-dose tacrolimus OD and mycophenolic acid. Group 2 will be treated with Basiliximab induction followed by standard-dose tacrolimus OD, mycophenolic acid and steroids. Group 3 will be treated with basiliximab induction followed by standard-dose tacrolimus OD for six months, whereafter the dose will be reduced plus mycophenolic acid and steroids. The total study period will be 2 years. Primary endpoint will be renal function, proteinuria and microalbuminuria measured 24 months after transplantation. Renal function will be measured by serum Creatinine, Creatinine clearances and CKD-EPI. Secondary endpoints will be the degree of tubular atrophy and interstitial fibrosis and the degree of arteriolar hyalinosis in renal biopsies taken at 12 and 24 months after transplantation. Biopsies will be evaluated according to the Banff Criteria for Renal Allograft Biopsy Interpretation. Quantitative morphometric analysis of interstitial fibrous tissue will be performed using the digital image analysis technique. Other secondary endpoints are patient and graft survival, the incidence of allograft rejection, cardiovascular accidents, pulse wave velocity, blood pressure, the number of antihypertensives, lipid profile, the incidence of malignancies, the incidence of infectious complications, the incidence of post transplant diabetes mellitus and the development of osteoporosis.

ELIGIBILITY:
Inclusion Criteria:

* recipient of a kidney graft (first of second) from a deceased or living (non-HLA identical) donor

Exclusion Criteria:

* patients with multi-organ transplants
* patients who are receiving a third or fourth transplant
* patients who have > 75% (current of historic) panel reactive antibodies
* patients receiving a kidney from a HLA identical living donr
* female patients who are pregnant or unwilling to used adequate contraception during the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2011-04; Primary Completion 2015-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
renal function parameters | 24 months
  renal function as measured by serum Creatinine and Creatinine Clearance, CKD-EPI, proteinuria

SECONDARY OUTCOMES:
tubular atrophy and interstitial fibrosis | 24 months
  tubular atrophy and interstitial fibrosis in renal biopsies
rejection episodes | two years
  number of treated biopsy proven acute rejection episodes (as scored by pathologist via Banff classification)
graft and patient survival | two years
  graft and patient survival
myocardial infarctions | two years
  number of myocardial infarctions
cerebrovascular accidents | two years
  number of cerebrovascular accidents
number of participants with infectious complications | two years
  bacterial and viral infections as measured by culture (bacterial infections) or PCR (viral infections)
number of participants with osteoporosis | 2 years
  as established by dexa bone densitometry

CONTACTS AND LOCATIONS:
Overall Officials: Jan-Stephan Sanders, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (3):
- Netherlands (3):
  - Academisch Medisch Centrum, Amsterdam
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden

REFERENCES:
- [Derived] van den Born JC, Meziyerh S, Vart P, Bakker SJL, Berger SP, Florquin S, de Fijter JW, Gomes-Neto AW, Idu MM, Pol RA, Roelen DL, van Sandwijk MS, de Vries DK, de Vries APJ, Bemelman FJ, Sanders JSF. Comparison of 2 Immunosuppression Minimization Strategies in Kidney Transplantation: The ALLEGRO Trial. Transplantation. 2024 Feb 1;108(2):556-566. doi: 10.1097/TP.0000000000004776. Epub 2024 Jan 19. PMID 37650722